CLINICAL TRIAL: NCT04777292
Title: A Randomized Controlled Trial of a Mobile Health Application for Enhancing Mental Health Literacy About Obsessive-compulsive Disorder and Reduce Stigmatizing Attitudes in Community (ESTOCMA)
Brief Title: ESTOCMA: Mental Health Application for Enhancing Mental Health Literacy About Obsessive-compulsive Disorder
Acronym: ESTOCMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Gemma García-Soriano, Associate professor, University of Valencia
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 29401; RTI2018-098349-B-I00 (Other Grant/Funding Number: ERDF/Ministry Science&Innovation,State Research Agency-Spain)
Record Dates: First submitted 2021-02-23; First posted 2021-03-02 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: mental health literacy; randomized controlled trial; obsessive-compulsive disorder; stigma; seeking help
MeSH Terms: conditions — Obsessive-Compulsive Disorder; Social Stigma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate-use (Experimental): Immediate use of esTOCma mobile app. Participants will use the mobile application immediately after the baseline assessment (T0) during approximately 10 days or until app completion.
  Interventions: Device: Use of a mobile health application until app completion
- Delayed use (Active Comparator): Delayed use of esTOCma mobile app. Participants will start using the app 10 days after the first assessment (T0), and immediately after the T1 assessment.
  Interventions: Device: Use of a mobile health application until app completion

INTERVENTIONS:
Device: Use of a mobile health application until app completion — Participants are asked to use esTOCma app approximately during 10 days, until app completion. This app has been designed to increase knowledge about obsessive-compulsive disorder (OCD), help seeking attitudes, and reduce stigmatizing attitudes. It consists in a game in which participants are asked to fight against the OCD stigma monster through ten missions. Participants have to liberate 10 characters who are prisoners of EsTOCma monster.
  Other Names: Use of esTOCma app

SUMMARY:
The aim of the study is to analyze the efficacy of a mobile health application (app) designed to increase mental health literacy, help seeking attitudes and reduce stigma associated with obsessive-compulsive disorder. A randomized controlled trial with crossover design will be carried out in non-clinical population to assess pre-post changes in levels mental health literacy, help seeking attitudes and stigma through app completion (an estimation of 10 days). Moreover, the stability of the changes will be tested at 3 months. Participants from community will be randomly assigned to one of two conditions: undertaking immediate-use or delayed use. We hypothesized that after using the app, participants will have a greater knowledge about obsessive-compulsive disorder, will be more prone to ask for help in case of showing OCD symptoms, and will show lower stigma attitudes and social distance.

DETAILED DESCRIPTION:
Stigmatizing attitudes are a problem associated to mental disorders. In obsessive-compulsive disorder (OCD) stigma has been associated to shame, guilty and delay asking for help. The aim of the study is to analyze the efficacy of a mobile health application (app) designed to increase mental health literacy, help seeking attitudes and reduce stigma associated with obsessive-compulsive disorder. The app has been named esTOCma. It consists in a game in which participants are asked to fight against the OCD stigma monster through ten missions. Participants have to liberate 10 characters who are prisoners of EsTOCma monster. A randomized controlled trial with crossover design will be carried out in non-clinical population to assess pre-post changes in levels mental health literacy, help seeking attitudes and stigma through app completion. Participants from community will be randomly assigned to one of two conditions: undertaking immediate-use (experimental group) or delayed-use (wait list control group) of the intervention through the esTOCma mobile app. Participants will be randomized through the app either to the experimental or control group. Then, within each group, participants will be randomized to one of six vignettes describing different obsessive-compulsive contents, and will be asked to complete baseline questionnaires (T0). Participants in the experimental group will be allowed to start using the app immediately after completing T0 and until completing the game (approximately 10 days). Immediately after finishing the app they will be asked to complete the post intervention assessment (T1), and then, 10 days after they will be asked to complete a follow up (T2). Participants in the control group will work as a waiting list comparison, in this sense, after completing the baseline assessment (T0), they will not be allowed to use the app. Then, days after completing the baseline questionnaires will be asked to complete again the baseline assessment (T1), and then, they will be allowed to begin the game until completing it. After, they will be asked to complete the post intervention assessment (T2). All participants will be asked to complete again the questionnaires 3 months after the post intervention assessment.

ELIGIBILITY:
Inclusion Criteria:

* having 18 years old or more
* mobile phone

Exclusion Criteria:

- having an obsessive-compulsive disorder diagnosis or suspictious of having OCD

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 228 (Actual)
Dates: Start 2021-12-21 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
Change in mental health literacy about obsessive-compulsive disorder | Through app completion, an average 10 days, and at 3 months follow-up
  Score change in mental health literacy (MHL) from baseline to app completion. MHL will be assessed through a self-report questionnaire developed ad hoc to assess general OCD knowledge and OCD identification. It is composed by 8 items with different alternatives. Correct answers will be computed. Higher score indicates higher number of correct answers, that is, higher OCD knowledge and identification.
Change in stigmatizing attitudes associated with obsessive-compulsive disorder | Through app completion, an average 10 days, and at 3 months follow-up.
  Score change in stigma from baseline to app completion. Stigma will be assessed by the Spanish Mental Illness Stigma Attribution Questionnaire. It is composed by 27 items and a Likert scale from 1 to 9. Higher scores indicate higher stigmatizing attitudes.
Change in social distance associated with obsessive-compulsive disorder | Through app completion, an average 10 days, and at 3 months follow-up.
  Score change in social distance from baseline to app completion. Social distance will be measured through a self-report questionnaire: Social Distance Scale, 7 items, Likert scale from 0 to 3. Higher scores, higher social distance.
Change in help-seeking attitudes associated with obsessive-compulsive symptoms | Through app completion, an average 10 days, and at 3 months follow-up.
  Score change in attitudes toward seeking help from baseline to app completion. It will be assessed with a self-report questionnaire assessing intention of seeking from formal/ informal sources of help: the General Help Seeking Questionnaire. It is composed by 7 items with a Likert scale from 1 to 7. Higher scores indicate higher intentions of asking for help except in item 7 (reversed score).
Change in Obsessive-Compulsive symptoms | Through app completion, an average 10 days, and at 3 months follow-up
  Score change on distress caused by obsessive-compulsive symptoms from baseline to app completion.. It will be assessed with the Obsessive-Compulsive Inventory-Revised. It is an 18-item self-report questionnaire, rated on a 4-point scale ranging from 1 ("not at all") to 4 ("extremely") that provides a total score (ranging from 0 to 72) and scores on six subscales: washing, checking, ordering, obsessing, hoarding and neutralizing. The total score will be used.

SECONDARY OUTCOMES:
Change in Self-esteem | Through app completion, an average 10 days, and at 3 months follow-up
  Score change in self-esteem from baseline to app completion. It will be assessed with the Single-Item Self-esteem Scale, a single item to measure self-esteem (i.e., I have high self-esteem) on a 5-point Likert Scale ranging from 1 ("not very true of me") to 5 ("very true of me"). The scale has strong convergent validity with the Rosenberg Self-Esteem Scale and showed similar predictive validity.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Valencia/ Universitat de València, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chaves A, Arnaez S, Castilla D, Roncero M, Garcia-Soriano G. Enhancing mental health literacy in obsessive-compulsive disorder and reducing stigma via smartphone: A randomized controlled trial protocol. Internet Interv. 2022 Jul 13;29:100560. doi: 10.1016/j.invent.2022.100560. eCollection 2022 Sep. PMID 35874968
- [Derived] Garcia-Soriano G, Arnaez S, Chaves A, Del Valle G, Roncero M, Moritz S. Can an app increase health literacy and reduce the stigma associated with obsessive-compulsive disorder? A crossover randomized controlled trial. J Affect Disord. 2024 Apr 1;350:636-647. doi: 10.1016/j.jad.2024.01.168. Epub 2024 Jan 20. PMID 38253133